CLINICAL TRIAL: NCT05320705
Title: The Effect of Intra Operative Dexmedetomidine in Prevention of Early Postoperative Atrial Fibrillation in Patients Undergoing Thoracic Non Cardiac Surgeries: a Randomized Controlled Trial
Brief Title: The Effect of Intra Operative Dexmedetomidine in Prevention of Early Postoperative Atrial Fibrillation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-17-2022
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer generated numbers and concealed by serially numbered, opaque and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelopes will be opened by the nurse, the card inside will determine the patient group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dexmedetomidine (Active Comparator): dexmedetomidine will be administered as a bolus dose, before the surgical incision, followed by infusion and stopped at the end of operation
  Interventions: Drug: Intra Operative Dexmedetomidine
- normal saline placebo (Placebo Comparator): similar bolus and infusion volumes of normal saline will be administered
  Interventions: Drug: Intra Operative Dexmedetomidine

INTERVENTIONS:
Drug: Intra Operative Dexmedetomidine — Dexmedetomidine will be administered as a bolus dose, before the surgical incision with 1mcg/kg iv in 100 ml saline solution over 10 minutes followed by infusion rate of 0.5 μg/kg per h infusion via syringe pump during surgery and stopped at the end of operation. Similar bolus and infusion volumes of normal saline will be administered in the Control group (placebo) However, anaesthesiologists will be permitted to reduce dose of the study drug as necessary to preserve haemodynamic stability.
  Other Names: intra operative precedex

SUMMARY:
The incidence of atrial fibrillation (AF) after lung resection varies between 12% and 30% after lobectomy and 23%-67% after pneumonectomy. The average time of onset of AF after lung resection is 2-3 days. AF after pulmonary resection can cause symptoms, hemodynamic instability, and stroke.Furthermore, AF following pulmonary resection may triple the mean duration stay in the intensive care unit and increase the total length of hospital stay by 2-9 days, with an increased in associated hospitalization costs.lastly, AF after lung resection has been associated with an increased risk of mortality , although the arrhythmia is more likely to be a consequence of other associated cardiopulmonary complications, rather than the main cause of death.

our study aim to assess the role of intra operative dexmedetomidine in reduction of early postoperative atrial fibrillation in patients undergoing thoracic non cardiac surgeries.

Objectives:

1. To evaluate possible efficacy of intraoperative dexmedetomidine in reduction of postoperative atrial fibrillation in patients undergoing thoracic non cardiac surgeries
2. To determine the incidence of new-onset atrial fibrillation after thoracic non cardiac surgeries in patients given intra operative dexmedetomidine

DETAILED DESCRIPTION:
This a randomized control trial is designed to include (350) patients ASA physical status II patients ranging from(18) to(70)years old scheduled for thoracic non cardiac surgeries

Patients meeting the inclusion criteria will be randomly assigned to receive either :

Group I : dexmedetomidine: (n=175) dexmedetomidine will be administered as a bolus dose, before the surgical incision with 1mcg/kg iv over 10 minutes followed by infusion rate of 0.5 μg/kg per h and stopped at the end of operation.

GroupII: normal saline placebo:(n=175) similar bolus and infusion volumes of normal saline will be administered as dexmedetomidine group

Anesthesia management

Preoperative procedures:

Full history and investigation will be taken in the form of CBC, blood sugar ,liver function tests. Kidney function tests ,electrolytes and coagulation profile Preoperative awake supine trans thoracic echocardiograms will be performed before operation using a 2.5/2.0- MHz transducer for imaging and Doppler echocardiography. Preoperative 12-leads will be performed to all patients. On arrival of the patient to the operating theatre and before induction of anesthesia, all standard monitors will be applied, including heart rate (HR), ECG, oxygen saturation (SpO2), end-tidal CO2, arterial blood pressure (systolic, diastolic, and MAP), and temperature, arterial catheter will be inserted in the radial artery for continuous blood pressure monitoring and frequent blood gas analysis. Initial readings of all these monitors will be taken and recorded before starting any drug infusion. After securing IV access by 20G cannula, all patients will be premedicated with 0.05mg/kg midazolam for anxiety, antibiotic 50mg/kg.

Intraoperative procedures:

Induction of general anesthesia will be done by fentanyl 2ug/kg/ iv, 2mg \kg propofol, and 0.5mg\kg atracurium to facilitate endotracheal intubation. Anesthesia maintenance will be achieved with endotracheal tube with suitable size, 1.2 minimum alveolar concentration of isoflurane, volume controlled mode ventilation, respiratory rate will be adjusted according to Et CO2 to range between 35-40 mmHg, a tidal volume of 6-8 ml/kg and mixture of gases in proportion 50% oxygen and 50% air, with PEEP 5 cm H2O and0.1 mg\kg atracurium every 30 min.10mg morphine intravenous will be given after induction and intubation.

Intervention Dexmedetomidine will be administered as a bolus dose, before the surgical incision with 1mcg/kg iv in 100 ml saline solution over 10 minutes followed by infusion rate of 0.5 μg/kg per h infusion via syringe pump during surgery and stopped at the end of operation. Similar bolus and infusion volumes of normal saline will be administered in the Control group (placebo) However, anaesthesiologists will be permitted to reduce dose of the study drug as necessary to preserve haemodynamic stability(systolic blood pressure decrease more than 20% from the baseline or\ and heart rate less than 60 ). with occurence of bradycardia and \or hypotension it will be managed by the attending anesthesiologist according to standard institutional guidelines and drug infusion rate will be decreased to the half. if bradycardia or hypotension persisted, drug infusion will be unblinded, stopped and reported as a serious side effect occured with drug infusion .By the end of surgery, anaesthesia will be discontinued ,patient will be reversed by neostigmine 0.05mg\kg and atropine0.02mg\kg, extubation will be done and patient will be transferred to post anaesthesia care unit (PACU).

Postoperative

1. Postoperative analgesia will be started with continuous infusion of 30 mg morphine associated with 180 mg ketorolac in 250 ml of normal saline at 5 ml /h and paracetamol infusion 1 g every 6 h. Additional bolus dose of 0.04mg/kg if vas exceed or equal 4 and it will be repeated if pain exist every 6 hours. All patients will be continuously monitored by 5-leads ECG and pulse oximeter(oxygen saturation) .12-leads ECG will be performed in occurence of tachycardia or arrythmia for the first 72 hours. Diagnoses of atrial fibrillation in the cardiac ICU will be made by clinicians who will be masked to group allocation. Atrial fibrillation will be defined by: clinician diagnosis; documented arrhythmia lasting at least 5 min ( supraventricular tachyarrhythmia characterized by uncoordinated atrial activation .Electrocardiographic findings include the replacement of the normal consistent p waves with oscillatory or fibrillatory waves of different sizes amplitudes and timing with narrow QRS complex unless other conduction abnormalities exist ( e.g. bundle branch block , accessory pathways). The ventricular response is often rapid and between 90 and 170 beats per minute and it will be documented by 12- lead ECG.
2. Post operative haemodynamic will be assessed (heart rate , ,systolic and diastolic blood pressure every 2 hours or with the occurrence of dysrhythmia)
3. Serial cardiac enzymes concentration (CK MB , Troponin ) will be measured every 6 h to rule out myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Gender both males and females
2. ASA Class II
3. Age 18-70 years
4. Patients undergoing thoracic non cardiac surgeries(lobectomy, pneumonectomy, and esophagectomy).

Exclusion Criteria:

A. Hypersensitivity or known allergy to dexmedetomidine. b.Patients with Sick-sinus orWolff-Parkinson-White syndromes; atrioventricular block atrial fibrillation within 30 days; a permanent pacemaker; used amiodarone or dexmedetomidine within30 days.

c. Patients with echocardiographic finding of an ejection fraction <30% and left atrial diameter more than 45mm and use of beta blockers or statins.

d. Liver and renal impairment(elevated liver enzymes (ALT, AST two to three fold), CRF ) e .Emergency operations ,video assisted thoracic surgeries and operation for spontaneous pneumothorax

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of new onset early atrial fibrillation following thoracic non cardiac surgeries in the first 72 hours postoperative | it will be measured in the first 72 hours postoperative
  Diagnoses of atrial fibrillation in the cardiac ICU will be made by clinicians who will be masked to group allocation. Atrial fibrillation will be defined by: clinician diagnosis; documented arrhythmia lasting at least 5 min ( supraventricular tachyarrhythmia characterized by uncoordinated atrial activation .Electrocardiographic findings include the replacement of the normal consistent p waves with oscillatory or fibrillatory waves of different sizes amplitudes and timing with narrow QRS complex.The ventricular response is often rapid and between 90 and 170 beats per minute and it will be documented by 12- lead ECG.

SECONDARY OUTCOMES:
The incidence of Dexmedetomidine side effects in the first 72 hours postoperative | it will be measured in the first 72 hours postoperative
  (hypotension , nausea , vomiting, dry mouth , bradycardia (HR <60 beats/ min), pyrexia, chills, hyperglycemia, hypocalcemia and acidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed nabih, lecturer, Principal Investigator — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No